CLINICAL TRIAL: NCT00620074
Title: Phase IV Open-Label Pilot Study to Evaluate the Combination of Voriconazole and Anidulafungin for the Treatment of Subjects With Proven or Probable Invasive Aspergillosis Who Are Intolerant of Polyene Treatment
Brief Title: Study to Test the Combination of Voriconazole and Anidulafungin in Patients Who Have, or Are Thought to Have, Invasive Aspergillosis and Who Are Unable to Take a Common Antifungal Therapy (Polyene)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See Detailed Description
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A8851014
Record Dates: First submitted 2008-02-08; First posted 2008-02-21 (Estimated); Results first posted 2010-02-15 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-01

CONDITIONS: Aspergillosis
Keywords: invasive aspergillosis, opportunistic mold infection
MeSH Terms: conditions — Aspergillosis | interventions — Voriconazole; Anidulafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- combination 2 (Experimental): anidulafungin plus voriconazole
  Interventions: Drug: voriconazole
- combination 1 (Experimental): anidulafungin plus voriconazole
  Interventions: Drug: anidulafungin

INTERVENTIONS:
Drug: voriconazole — Subjects with creatinine clearance at least 50 ml/min will receive initial treatment with IV (loading dose of 6 mg/kg Q12h followed by maintenance dose of 4 mg/kg Q12h) or oral (loading dose of 400 mg Q12h followed by maintenance dose of 300 mg Q12h). Subjects with creatinine clearance <50 ml/min will receive oral voriconazole (loading dose of 400 mg Q12h followed by maintenance dose of 300 mg Q12h).
  Other Names: Vfend
  Arms: combination 2
Drug: anidulafungin — Loading dose of 200 mg QD followed by maintenance dose of 100 mg QD for up to a total of 28 days therapy
  Other Names: Eraxis
  Arms: combination 1

SUMMARY:
This study will test the effectiveness and the safety of giving two antifungal agents (voriconazole and anidulafungin) together to treat invasive aspergillosis in patients who are unable to tolerate polyene therapy.

DETAILED DESCRIPTION:
The study was terminated on January 12, 2009 due to the overall low rate of enrollment. The decision to terminate the trial was not based on any safety concerns. Patients who were enrolled in the study prior to January 12, 2009 were allowed to remain in the study until completing their participation as specified in the protocol.

ELIGIBILITY:
Inclusion Criteria:

Proven or probable invasive aspergillosis. Patient is intolerant to polyene therapy.

Exclusion Criteria:

Patients with invasive aspergillosis for more than 30 days at the time of study entry. Patients with uncontrolled bacterial or viral infection at the time of study entry. Patients with significant liver dysfunction or who are taking certain medications which interact with voriconazole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Fort Worth, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8851014&StudyName=Study%20to%20Test%20the%20Combination%20of%20Voriconazole%20and%20Anidulafungin%20in%20Patients%20Who%20Have%2C%20or%20are%20Thought%20to%20Have%2C%20Invasive%20Aspergillosis

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was closed due to an overall low rate of enrollment after only 6 subjects enrolled.
Groups:
- Anidulalfungin and Voriconazole: Voriconazole: subjects with creatinine clearance at least 50 milliliters per minute (ml/min) will receive initial treatment with intravenous (IV) (loading dose of 6 milligrams per kilogram [mg/kg] every 12 hours [Q12h]) followed by maintenance dose of 4 mg/kg Q12h or oral (PO) (loading dose of 400 mg Q12h followed by maintenance dose of 300 mg Q12h). Subjects with creatinine clearance <50 ml/min will receive oral Voriconazole (loading dose of 400 mg Q12h followed by maintenance dose of 300 mg Q12h).
  Anidulafungin: loading dose of 200 mg once daily (QD) followed by maintenance dose of 100 mg QD for up to a total of 28 days therapy.
  Subjects remain on combination therapy for minimum of 14 days and a maximum of 28 days; after combination therapy complete, subjects may remain on a maintenance dose of Voriconazole monotherapy until Day 42.
Period: Overall Study
Arm/Group | Anidulalfungin and Voriconazole
Started | 6
Completed | 5
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Anidulalfungin and Voriconazole
Number analyzed (Participants) | 6
Age, Customized [Number; unit: participants]
  Between 57 and 83 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Summary of Global Response at End of Treatment (EOT)
Description: Number of subjects with global response consisting of a combination of clinical and radiological findings at the end of therapy. Possible outcome categories: Complete Response: resolution of all clinical signs and symptoms and more than 90% of lesions due to invasive aspergillosis that were visible on radiological studies; Partial Response: clinical improvement and greater than 50% improvement in radiological findings; Stable Response: no change from baseline or an improvement of less than 50% in radiological findings; Failure (no response): worsening disease.
Time Frame: End of Treatment (Day 42)
Population: Intent-to-treat (ITT): includes all subjects who received at least 1 dose of study medication. No descriptive or inferential analysis was completed due to low enrollment and subsequent early termination of study.
Measure: Number; unit: participants
Groups:
- Anidulalfungin and Voriconazole: Anidulafungin and voriconazole in combination followed by monotherapy.
Arm/Group | Anidulalfungin and Voriconazole
Number analyzed (Participants) | 6
participants
  Failure (No response) | 1
  Partial response | 3
  Stable response | 0
  Complete response | 2

2. Secondary Outcome: Summary of Global Response at Week 2, Week 4, and Week 6
Description: as for outcome 1
Time Frame: Week 2, Week 4, Week 6
Population: ITT; due to low study enrollment, data not summarized by global response at Week 2, Week 4, and Week 6. Cross-reference outcome measure: Summary of Global Response at End of Treatment (EOT).
Measure: Number; unit: participants
Arm/Group | Anidulalfungin and Voriconazole
Number analyzed (Participants) | 0

3. Secondary Outcome: Summary of Mortality
Description: Number of subects with documented mortality (death).
Time Frame: Up to Week 6
Population: ITT
Measure: Number; unit: participants
Arm/Group | Anidulalfungin and Voriconazole
Number analyzed (Participants) | 6
participants | 1

4. Secondary Outcome: Galactomannan Titer Assay Levels and Global Response
Description: Number of subjects per Galactomannan titer level with global response for all subjects (with or without renal impairment). The galactomann assay is an immunological blood serum test used to diagnose invasive aspergillosis and to monitor disease progression. Global response is a composite of clinical and radiological findings summarized as Complete Response: resolution of all clinical signs and symptoms; Partial Response: clinical improvement; Stable Response: no change from baseline or an improvement of less than 50% in radiological findings; Failure (no response): worsening disease.
Time Frame: Up to Week 6
Population: ITT. No descriptive or inferential analysis was completed due to low enrollment and subsequent early termination of study.
Measure: Number; unit: participants
Arm/Group | Anidulalfungin and Voriconazole
Number analyzed (Participants) | 0

5. Secondary Outcome: Voriconazole Trough Levels With Intravenous and Oral Dosing
Description: Voriconazole trough plasma concentrations measured as nanograms per milliliter (ng/mL).
Time Frame: Week 1 through Week 6
Population: ITT; only 1 pharmacokinetic sample was collected for each subject, therefore a comprehensive analysis of trough plasma concentrations was not completed due to insufficient data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Anidulalfungin and Voriconazole
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Anidulalfungin and Voriconazole
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulalfungin and Voriconazole (N=6)
Disease progression (General disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulalfungin and Voriconazole (N=6)
Anaemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 1
Oropharyngeal candidiasis (Infections and infestations) | 1
Blood glucose increased (Investigations) | 1
Blood magnesium decreased (Investigations) | 1
Blood potassium increased (Investigations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Metabolic alkalosis (Metabolism and nutrition disorders) | 1
Anxiety (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Subclavian vein thrombosis (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Due to low enrollment and early termination of the study, data was insufficient for descriptive or inferential analysis as planned; no significant treatment-related safety results were identified in the subjects treated with combination therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.